CLINICAL TRIAL: NCT00002273
Title: Double-Blind, Placebo-Controlled Study of Intravenous Ganciclovir (DHPG) for Cytomegalovirus Colitis in Patients With Acquired Immune Deficiency Syndrome
Brief Title: A Study of Ganciclovir in the Treatment of Cytomegalovirus of the Large Intestine in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 029C; ICM 1288
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-09

CONDITIONS: Colitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Cytomegalovirus Infections; Colitis; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Colitis; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To attempt to demonstrate the efficacy of ganciclovir (DHPG) treatment of cytomegalovirus (CMV) colitis in AIDS patients by evaluating both clinical and virologic parameters. To determine acceptability and the safety profile of a 2-week course of intravenous (IV) DHPG therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* An underlying diagnosis of AIDS by CDC surveillance definition (group IV, category c-1 or subgroup D only).
* Colitis manifested clinically by diarrhea.
* Colon biopsy demonstrating a typical histologic picture of cytomegalovirus (CMV) disease.
* Cultures for CMV from blood and urine should be obtained within 1 week of study entry but need not be positive prior to entry. (A positive culture is needed for final inclusion in AN.)

Prior Medication:

Allowed:

* Topical acyclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* History of chronic or acute liver disease.
* History of significant mental illness.
* Life expectancy < 1 month.
* Presence of any cause of colitis other than cytomegalovirus (CMV). (The following tests must be negative:
* Stool culture for enteric bacterial pathogens, stool exam for ova and parasites, stool exam for cryptosporidia, stool exam for AFB.) Colitis that is so severe that it would be against the patient's best interest to be treated with placebo for 2 weeks prior to being eligible to receive ganciclovir (DHPG) on a "compassionate" use basis. Patients with a colitis of this severity should be treated with DHPG on "compassionate" use basis.
* Presence of clinically significant extra-colonic active CMV disease of retina or visceral organs (which could progress during the no-treatment period).
* Presence of significant renal disease resulting in any decrement of creatinine clearance from normal.

Concurrent Medication:

Excluded:

* Any other investigational drug, whether or not as part of a formal clinical study.

Patients with the following are excluded:

* History of chronic or acute liver disease.
* History of significant mental illness.
* Life expectancy < 1 month.
* Presence of any cause of colitis other than cytomegalovirus (CMV). (The following tests must be negative:
* Stool culture for enteric bacterial pathogens, stool exam for ova and parasites, stool exam for cryptosporidia, stool exam for AFB.) Colitis that is so severe that it would be against the patient's best interest to be treated with placebo for 2 weeks prior to being eligible to receive ganciclovir (DHPG) on a "compassionate" use basis. Patients with a colitis of this severity should be treated with DHPG on "compassionate" use basis.
* Presence of clinically significant extra-colonic active CMV disease of retina or visceral organs (which could progress during the no-treatment period).
* Presence of significant renal disease resulting in any decrement of creatinine clearance from normal.

Prior Medication:

Excluded within 2 days of study entry:

* Nucleoside analogs.
* Excluded within 1 week of study entry:
* Antimetabolites or interferon.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Roche Global Development - Palo Alto, Palo Alto, California, United States

REFERENCES:
- [Background] Dieterich DT, Kotler DP, Busch DF, Crumpacker C, Du Mond C, Dearmand B, Buhles W. Ganciclovir treatment of cytomegalovirus colitis in AIDS: a randomized, double-blind, placebo-controlled multicenter study. J Infect Dis. 1993 Feb;167(2):278-82. doi: 10.1093/infdis/167.2.278. PMID 8380610